CLINICAL TRIAL: NCT01343576
Title: Effect of Dairy Fat on Plasma Phytanic Acid in Healthy Volunteers - A Randomized Controlled Study
Brief Title: Effect of Dairy Fat on Plasma Phytanic Acid in Human
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Collaborators: The Danish Dairy Research Foundation, Denmark (Other); The Danish Council for Strategic Research (Other)
Responsible Party: Tine Tholstrup, Dpt Human Nutrition, University of Copenhagen, Denmark
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: H-B-2009-052 (Adel)
Record Dates: First submitted 2011-04-18; First posted 2011-04-28 (Estimated); Last update posted 2011-04-28 (Estimated); Status verified 2009-11

CONDITIONS: Coronary Heart Disease
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Dietary Supplement: milk fat — 45 g milk fat per day in 4 weeks
  Other Names: yellow group; Green group

SUMMARY:
The aim of the study is to investigate if cow feeding regimes affects concentration of plasma phytanic acid and risk markers of the metabolic syndrome in human.

ELIGIBILITY:
Inclusion Criteria:

* sign written consent
* Age: 20-42
* BMI: 20-30
* increased risk of developing MS
* refrain from dietary supplements and blood donations prior to, and during the study

Exclusion Criteria:

* poor compliance
* if they suffering from any chronic or long lasting illness
* abuse of alcohol or medicine

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2009-08; Primary Completion 2009-11 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
plasma phytanic acid | before and after the intervention (4 weeks)

SECONDARY OUTCOMES:
total cholesterol | before and after the intervention (4 weeks)
LDL cholesterol | before and after the intervention (4 weeks)
HDL cholesterol | before and after the intervention (4 weeks)
triacylglycerol | before and after the intervention (4 weeks)
C-reactive protein | before and after the intervention (4 weeks)
insulin | before and after the intervention (4 weeks)
glucose | before and after the intervention (4 weeks)
fatty acid composition in plasma | before and after the intervention (4 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Tine Tholstrup, lector, Principal Investigator — Department of Human Nutrition, University of Copenhagen
Locations (1):
- Department of Human Nutrition, Frederiksberg, Denmark

REFERENCES:
- [Derived] Werner LB, Hellgren LI, Raff M, Jensen SK, Petersen RA, Drachmann T, Tholstrup T. Effect of dairy fat on plasma phytanic acid in healthy volunteers - a randomized controlled study. Lipids Health Dis. 2011 Jun 10;10:95. doi: 10.1186/1476-511X-10-95. PMID 21663648